CLINICAL TRIAL: NCT06991647
Title: Effectiveness of Adjuvant Premedication of Intranasal Dexmedetomidine on the Intubation Procedure in Children
Brief Title: Effectiveness of Intranasal Dexmedetomidine Premedication in Child Intubation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Raihanita Zahra, Clinical Research Coordinator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-09-1444
Record Dates: First submitted 2025-05-05; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Elective Surgical Procedure; ASA Physical Status I; ASA Physical Status II
Keywords: intranasal dexmedetomidine
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive 1 ml of 0.9% NaCl solution administered intranasally using a 1 ml syringe connected to a nasal device.
  Interventions: Drug: 0.9% NaCl solution
- Intranasal dexmedetomidine (Experimental): Participants will receive intranasal dexmedetomidine at a dose of 2 mcg/kg body weight, diluted in 1 mL of 0.9% NaCl, administered using a 1 mL syringe connected to a nasal device.
  Interventions: Drug: Intranasal dexmedetomidine

INTERVENTIONS:
Drug: Intranasal dexmedetomidine — Intranasal dexmedetomidine at a dose of 2 mcg/kg body weight, diluted in 1 mL of 0.9% NaCl, administered using a 1 mL syringe connected to a Teleflex MAD Nasal device while in the supine position. The soft tip of the device will be gently placed into each nostril without applying pressure. The solution will be sprayed slowly to create a fine mist. The total dose will be divided equally, with 0.5 mL delivered into each nostril, administered approximately 30 minutes before intubation during induction.
  Arms: Intranasal dexmedetomidine
Drug: 0.9% NaCl solution — Participants will receive 1 ml of 0.9% NaCl solution administered intranasally using a 1 ml syringe connected to a Teleflex MAD nasal device while in the supine position. The soft tip of the Teleflex MAD nasal device is gently placed into each nostril without applying pressure. The solution is slowly sprayed to create a fine mist for patient comfort. The dose is divided equally, delivering 0.5 ml into each nostril, approximately 30 minutes before intubation during induction.
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out if a medicine called dexmedetomidine, given as a nasal spray, can help patients stay calm and comfortable before having a breathing tube placed (intubation). Researchers want to see if using this nasal spray affects blood pressure, heart rate, comfort with the oxygen mask, how quickly the tube is placed, and how sleepy patients become. They also want to check if patients who receive dexmedetomidine need less pain medicine (Fentanyl) during the procedure. Participants will receive either the dexmedetomidine nasal spray or a plain saltwater spray (placebo). Doctors will then measure blood pressure, heart rate, comfort levels, time needed for intubation, sleepiness, and the amount of pain medication used.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-6 years undergoing elective surgery
* ASA physical status 1 and 2

Exclusion Criteria:

* Children with difficult airway
* Active infection in nasal and oral area
* Subjects with mental retardation, ADHD, and cerebral palsy
* Difficult intravenous access

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Mean arterial pressure | immediately before premedication and immediately after intubation
  Measured by non-invasive blood pressure monitoring
Heart rate | immediately before premedication and immediately after intubation
  Measured by electrocardiography electrodes in vital sign monitor
Mask acceptance | Before induction
  Measured using the Pediatric Anesthesia Behavior (PAB) scale. The PAB scale range from 1 to 3, with 1 indicating the best outcome (happy) and 3 the worst outcome (mad).
Intubation duration | during intubation
  Measured using stopwatch, in seconds Started when inserting laryngoscope into the mouth, ended when end tidal CO2 is detected by the monitor
Sedation Score | Immediately upon arrival to the operating room, before induction of anesthesia
  Sedation level was assessed using the COMFORT Behaviour Scale, which evaluates the child's sedation state after administration of dexmedetomidine. The total score ranges from 6 to 30, with the following interpretations:
  * Excessive sedation: 6-10
  * Adequate sedation: 11-22
  * Inadequate sedation: 23-30 Higher scores indicate less effective sedation control, whereas lower scores reflect deeper sedation.
Opioid use | Immediately after intubation
  Amount of fentanyl (per kg body weight) used during intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No